CLINICAL TRIAL: NCT02792322
Title: A Pilot Study Assessing Robotic Surgery in the Seated or Supine Position for Benign and Malignant Lesions of the Head and Neck Using the da Vinci Robotic Surgical Systems and Modified Transoral Instrumentation
Brief Title: Robotic Surgery in the Seated Position for Benign and Malignant Lesions of the Head and Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kathryn (Katie) M. Van Abel, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-001297; NCI-2022-10968 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-05-19; First posted 2016-06-07 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2024-08

CONDITIONS: Oropharyngeal Neoplasms; Head and Neck Cancer
Keywords: Cancer; Oropharynx
MeSH Terms: conditions — Oropharyngeal Neoplasms; Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trans Oral Robotic Surgery (TORS) (Other): Patient's are having TORS surgery in a seated position
  Interventions: Device: Transoral Robotic Surgery (TORS) with the daVinci Robotic Surgical System device

INTERVENTIONS:
Device: Transoral Robotic Surgery (TORS) with the daVinci Robotic Surgical System device — Patient's will be having TORS surgery in a seated position
  Other Names: Da Vinci Robotic Surgical Systems

SUMMARY:
This study is designed to investigate if transoral surgery with the patient in the seated position utilizing the da Vinci® Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) will enable better visualization and expedited removal of benign and malignant tumors of the throat.

DETAILED DESCRIPTION:
The da Vinci Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) being evaluated in this pilot study consists of 3 basic components: a surgeon's console, articulated mechanical arms and sterilizable instruments. The console includes a computer, video monitor and instrument controls, and is located in the operating room adjacent to the operating room table. The console is connected via computer to the mechanical arms holding the endoscope (surgical TV camera) and sterile surgical tools (e.g., forceps, scissors, electrocautery, etc.). These arms are located immediately adjacent to the patient on the operating room table. The surgeon sits at the console and controls the position and movement of the arms and surgical tools. The design of these tools is based upon well-established, commonly used surgical instruments. The da Vinci Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) is a "manual image-guided surgery" system that is computer enhanced rather than "computer guided robotic surgery" in which the surgeon programs the computer to do the surgery and the robot does the surgery (also known as a "milling" device). Use of the da Vinci Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) in the aforementioned configuration in fact facilitates an exact translation of the surgeon's hand and finger movements at the console to precise and tremor-free movements of the arms and instruments.

ELIGIBILITY:
Inclusion Criteria:

* Patient must present with indications for diagnostic or therapeutic surgery for benign or malignant diseases of the head and neck.
* Written informed consent.

Pre-Operative Exclusion Criteria:

* Unexplained fever and/or untreated, active infection.
* Patient pregnancy.
* Previous head and neck surgery precluding robotic procedures.
* The presence of medical conditions contraindicating general anesthesia or standard surgical approaches.

Intra-Operative Exclusion Criteria:

* It is recognized that sometimes patients cannot be excluded from study participation until prepped in the surgical suite such that their anatomy is exposed and available for medical analysis. The following situations represent instances whereby which patients would be excluded from this study based upon anatomical findings not evident in the pre-operative setting:
* Inability to adequately visualize anatomy or place robotic instrumentation to perform the diagnostic or therapeutic surgical approach in the seated position.
* In this circumstance, the procedure would be completed by standard robotic transoral surgery or an alternative approach may be chosen.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
TORS surgery completion in the seated position | Measures assessed at time of intervention (during surgery)
  Recording how many participants' surgery was completed in the seated position

SECONDARY OUTCOMES:
Length of participants' surgical time | Measures assessed at time of intervention (during surgery)
  Surgical start and stop times are recorded in the medical record
Estimated amount of blood loss during participants' surgery | Measures assessed at time of intervention (during surgery)
  Record blood loss during surgery as estimated by the lead surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Van Abel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holzgreve W, Miny P, Holzgreve A, Rehder H. [Ultrasound findings as a sign of fetal triploidy]. Ultraschall Med. 1986 Aug;7(4):169-71. doi: 10.1055/s-2007-1011939. German. PMID 3538408
- [Background] Weinstein GS, O'Malley BW Jr, Magnuson JS, Carroll WR, Olsen KD, Daio L, Moore EJ, Holsinger FC. Transoral robotic surgery: a multicenter study to assess feasibility, safety, and surgical margins. Laryngoscope. 2012 Aug;122(8):1701-7. doi: 10.1002/lary.23294. Epub 2012 Jul 2. PMID 22752997
- [Background] Matjasko J, Petrozza P, Cohen M, Steinberg P. Anesthesia and surgery in the seated position: analysis of 554 cases. Neurosurgery. 1985 Nov;17(5):695-702. doi: 10.1227/00006123-198511000-00001. PMID 4069324
- [Background] Engelhardt M, Folkers W, Brenke C, Scholz M, Harders A, Fidorra H, Schmieder K. Neurosurgical operations with the patient in sitting position: analysis of risk factors using transcranial Doppler sonography. Br J Anaesth. 2006 Apr;96(4):467-72. doi: 10.1093/bja/ael015. Epub 2006 Feb 7. PMID 16464980
- [Background] Van Abel KM, Moore EJ. The rise of transoral robotic surgery in the head and neck: emerging applications. Expert Rev Anticancer Ther. 2012 Mar;12(3):373-80. doi: 10.1586/era.12.7. PMID 22369328
- [Background] Moore EJ, Olsen KD, Martin EJ. Concurrent neck dissection and transoral robotic surgery. Laryngoscope. 2011 Mar;121(3):541-4. doi: 10.1002/lary.21435. Epub 2011 Jan 4. PMID 21344431
- [Background] Weinstein GS, O'Malley BW Jr, Desai SC, Quon H. Transoral robotic surgery: does the ends justify the means? Curr Opin Otolaryngol Head Neck Surg. 2009 Apr;17(2):126-31. doi: 10.1097/MOO.0b013e32832924f5. PMID 19342953
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials